CLINICAL TRIAL: NCT05370859
Title: Motivational Monitoring to Enhance Smoking Cessation Among Cancer Patients Pilot Study
Brief Title: mMe: Motivational Monitoring to Enhance Smoking Cessation Among Cancer Patients
Acronym: mMe
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kara Wiseman, MPH, PhD, Research Assistant Professor of Public Health Sciences, University of Virginia
Other Study IDs: 18184
Record Dates: First submitted 2022-04-27; First posted 2022-05-12 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Smoking Behaviors; Cancer; Motivation
MeSH Terms: conditions — Smoking; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mme Study Participants: Participants will complete a baseline survey, 11 weekly surveys, and a follow-up survey at 12 weeks
  Interventions: Other: There is no intervention for this study

INTERVENTIONS:
Other: There is no intervention for this study — There is no intervention or exposure for this study

SUMMARY:
The objectives of this study are to pilot test a protocol of weekly assessments of motivation to quit and other relevant constructs combined with information about how to enroll in cessation programs, which will allow initial quantification of motivation to quit during cancer treatment and develop hypotheses about the impact of motivation on the decision to enroll in services.

ELIGIBILITY:
Inclusion Criteria:

* An adult (18+)
* Current smoker defined by: Has smoked 100 cigarettes in their lifetime (may be multi-tobacco users as long as they also use combustible cigarettes).
* Any type of cancer (except non-melanoma skin cancer)
* Anticipates receiving any of the following cancer treatments in the 3 months following enrollment: chemotherapy, surgery, immunotherapy, bone marrow or stem cell transplant, hormone therapy, or radiation
* Access to the Internet

Exclusion Criteria:

* Not smoked 100 cigarettes in their lifetime
* < 18 years in age
* Diagnosed with non-melanoma skin cancer
* Not diagnosed with cancer
* Does not anticipate receiving cancer treatments in the 3 months following enrollment
* Has been previously enrolled in an existing Cancer Center Tobacco Treatment Program (TTP)
* Not comfortable reading and responding to questions in English
* No consistent access to the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being seen at the study recruitment sites for cancer treatment, who have a current cancer diagnosis and who are currently smoking. Other concurrent tobacco use is also acceptable.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Number of participants who enroll in cessation services | 12 weeks after study start
  Assessed using administrative records

SECONDARY OUTCOMES:
Level of and change in motivation and self-efficacy to quit smoking | Through study completion, an average of 12 weeks
  Assessed using self-report on the weekly and 12-week survey
Level of and change in anxiety and depression | Through study completion, an average of 12 weeks
  Assessed using self-report (PHQ-4) on the weekly and 12-week survey
Number of smoking quit attempts | 12 weeks after study start
  Assessed using self-report on the weekly and 12-week survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Cancer Center and affiliated sites, Charlottesville, Virginia, United States